CLINICAL TRIAL: NCT03837145
Title: Propofol for Sedation of Postoperative Electively Ventilated Liver Transplant Recipients-An Observational Study
Brief Title: Propofol for Sedation of Postoperative Electively Ventilated Liver Transplant Recipients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Rishabh Jaju, senior resident, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBS-TRANSPLANT ANESTHESIA-01
Record Dates: First submitted 2019-01-29; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Liver transplant recipients: Adult patients requiring elective post-operative ventilation after a living donor liver transplant receiving intravenous propofol infusion for sedation titrated to Bi-Spectral Index (BIS) score of 60-80,as per our institutional protocol.

SUMMARY:
All consenting, adult patients aged 18 years and above who will require elective ventilation after liver transplant recipient surgery will be enrolled for the study. Patients in acute liver failure, hepatic encephalopathy or patients with history of allergic reactions to propofol will be excluded from the study. This is an observational study. As per institute treatment protocol, propofol will be given post-operatively at a dose of 1 mg/kg/hr and than titrated to maintain a Bi-Spectral Index (BIS) score of 60-80 till the patient is on ventilator. There will be no deviation from our routine institutional protocol and no other sedative drugs like opioids or benzodiazepines will be used and no interventions will be done. Hemodynamics will be maintained targeting a mean arterial pressure (MAP) of at least 65 mm Hg. during the study period using appropriate measures.

ELIGIBILITY:
Inclusion Criteria:

• Living donor liver transplant (LDLT) recipient adult patients ≥ 18 years of age requiring postoperative elective ventilation.

Exclusion Criteria:

* Propofol allergy
* Acute liver failure (ALF).
* Hepatic encephalopathy (HE)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consenting LDLT recipient adult patients ≥ 18 years of age who require postoperative elective ventilation after recieving a living donor liver transplant.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Dosage of propofol in mg/kg/hr required for sedation (BIS:60-80) of postoperative electively ventilated living donor liver transplant recipients. | up to 24 hours
  Every 2 hrly , the continuous intravenous Propofol dose going on will be recorded.

SECONDARY OUTCOMES:
Changes of propofol dose over the study period to maintain BIS between 60 -80 | up to 24 hours
  Propofol doses will be recorded titrated to BIS of 60-80
Correlation of the mean dose of propofol in mg/kg/hr with Arterial ammonia at baseline and to see the association between immediate post operative and Postoperative day1 ammonia with corresponding propofol dose. | up to 24 hours
  Arterial ammonia levels will be noted pre-operatively, immediate post-operative and after extubation.
Correlation of propofol dose with respective arterial lactate levels every 2 hours during the period of elective ventilation | up to 24 hours
  Lactate levels will be recorded every 2 hrs till the patient is on ventilator

CONTACTS AND LOCATIONS:
Overall Officials: rishabh jaju, DNB, Principal Investigator — Institute of liver and biliary sciences,New Delhi-110070
Locations (1):
- Institute of liver and biliary sciences, New Delhi, National Capital Territory of Delhi, India